CLINICAL TRIAL: NCT02470416
Title: A Prospective Case Control Study on the Prevalence of Small Bowel and Colonic Polyps in Patients With Duodenal Adenomas/Ampullomas Who do Not Have Familial Adenomatous Polyposis (FAP) or Peutz Jeghers Syndrom (PJS).
Brief Title: Prevalence of Small Bowel Polyps in Patients With Sporadic Duodenal Adenomas
Acronym: SPIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Collaborators: Westmead hospital Westmead NSW 2145 Australia (Unknown)
Responsible Party: Principal Investigator, Professor Michael Bourke, Professor of medicine, Western Sydney Local Health District
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/14/WMEAD/226(4028)
Record Dates: First submitted 2015-06-02; First posted 2015-06-12 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Polyps
Keywords: duodenal; ampulla
MeSH Terms: conditions — Polyps | interventions — Endoscopy

ARMS (2):
- Case (Active Comparator): Patients who have had a previous diagnosis and/or treatment of a duodenal/ampullary polyp at Westmead hospital
  Interventions: Device: Small bowel video capsule endoscopy (VCE) GIVEN/COVIDIEN LTD
- Control (Active Comparator): Age matched controls having VCE for OGIB/IDA at Westmead hospital.
  Interventions: Device: Small bowel video capsule endoscopy (VCE) GIVEN/COVIDIEN LTD

INTERVENTIONS:
Device: Small bowel video capsule endoscopy (VCE) GIVEN/COVIDIEN LTD — Cases and controls will have a standard VCE procedure at our institution.

SUMMARY:
Little is known about the prevalence of small bowel polyps in patients with sporadic Duodenal/Ampullary polyps. The investigators aim to investigate the prevalence of small bowel polyps in patients with sporadic (ie not related to FAP or PJS) duodenal/ampullary adenomas by performing small bowel capsule endoscopy and comparing the results to those acquired from a control cohort undergoing VCE for accepted indication at our centre.

DETAILED DESCRIPTION:
Investigation for suspected SB tumors is an acceptable indication for VCE. SB polyps occur frequently in patients with FAP/PJS and in patients with FAP, they are significantly more common in patients with Duodenal/Ampullary polyps. Little is known about the prevalence of small bowel polyps in patients with sporadic Duodenal/Ampullary polyps.

The primary hypothesis is that patients with sporadic (ie not related to FAP or PJS) duodenal/ampullary adenomas have a higher prevalence of small bowel polyps compared with patients undergoing VCE for various indications who have not had a duodenal polyp diagnosed or removed.

Patients who have had a previous diagnosis and/or treatment of a duodenal/ampullary polyp at Westmead hospital will receive VCE examination. Control population will consist of age matched controls having VCE for OGIB/IDA at Westmead hospital. Patients will be required to have had a documented colonoscopy within the previous three years. If colonoscopy was not performed within this time frame, the patient will have a colonoscopy as part of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Cases - Patients who were diagnosed with or underwent resection of a duodenal adenoma/ampulloma at Westmead hospital between the years 2005-2014.
* Controls - Patients undergoing VCE procedure for the evaluation of obscure gastrointestinal bleeding (OGIB) or Iron deficiency anemia (IDA).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with sporadic (ie not related to FAP or PJS) duodenal/ampullary adenomas | 24 months

SECONDARY OUTCOMES:
Number of participants with presence and prevalence of colonic polyps | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, FRACP, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Awadie H, Klein A, Tate D, Jideh B, Bar-Yishai I, Goodrick K, Ahlenstiel G, Bourke MJ. The prevalence of small-bowel polyps on video capsule endoscopy in patients with sporadic duodenal or ampullary adenomas. Gastrointest Endosc. 2021 Mar;93(3):630-636. doi: 10.1016/j.gie.2020.07.029. Epub 2020 Jul 24. PMID 32717365